CLINICAL TRIAL: NCT05067569
Title: App-delivered Sleep ThERapy for Older Individuals With Insomnia (ASTEROID Study)
Brief Title: App-delivered Sleep ThERapy for Older Individuals With Insomnia
Acronym: ASTEROID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X21-0265
Record Dates: First submitted 2021-09-08; First posted 2021-10-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Insomnia
Keywords: sleep; digital; older people; brief behavioural therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be provided with a digital brief behavioural therapy (SleepFix app) which provides personalised sleep retraining therapy. Participants will also be provided a sleep-tracking wearable device (Fitbit) that synchronises the going to bed and getting out of bed times with the SleepFix app. Participants will complete a daily sleep diary and can modify the sleep-tracking wearable device sleep data. The program will provide an individualised sleep window of when to go and when to get out of bed. There are five stages focusing on bed timings, sleep efficiency and a maintenance phase for consolidating the new sleep pattern. The program provides information related to sleep hygiene and stimulus control. This will be available for participants for 6 weeks. An active wait-listed control of sleep health education will consist of 3 modules delivered biweekly of generalised sleep health information that could be found on the internet.
Who Masked: Investigator
Masking Description: Participants will not be blinded as they will know what treatment they receive. This is typical of behavioural interventions.
  Note: the study project coordinator will not be blinded as they will be managing the study such as sending sleep-tracking wearable devices to the intervention arm and communicating with participants. All investigators and data analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital brief behavioural therapy for insomnia (Experimental): Participants randomised to the digital brief behavioural therapy for insomnia (SleepFix app) will be provided an unique access code to download the app. The intervention uses sleep retraining therapy to reduce excess time spent in bed and retrain sleep by matching time in bed (minimum of five and a half hours) to total sleep time. All participants in the intervention arm will also be provided a sleep-tracking wearable device (Fitbit) which will synchronised bed times (going to bed and rising) and are synchronised with the SleepFix app. Participants wil complete a daily sleep diary, rate sleep quality and mood. The intervention is provided for 6 weeks.
  Interventions: Behavioral: SleepFix mobile application
- Sleep Health Education wait-list control (Active Comparator): Participants randomised to the control group will gain access to the first Sleep Health Education module immediately following completion of baseline questionnaires. There are three modules provided bi-weekly with information about sleep health and broad details about managing sleep disturbances. Participants will receive a link to this information as each module is made available.
  Upon completion of the study (week 26), the control group will receive free access to the SleepFix mobile application.
  Interventions: Behavioral: Sleep Health Education

INTERVENTIONS:
Behavioral: SleepFix mobile application — The SleepFix app is a novel, innovative way to deliver digital brief behavioural therapy for insomnia for adults.
  Arms: Digital brief behavioural therapy for insomnia
Behavioral: Sleep Health Education — These internet-based modules provide an active control intervention consisting of 3 modules provided bi-weekly. The participant will receive a link to this information as each module is made available. Control participants will have full access to these modules for the duration of the study. They reflect basic educational information regarding sleep health for poor sleepers that is otherwise easily accessible on the internet.
  Arms: Sleep Health Education wait-list control

SUMMARY:
This randomised, open, parallel controlled trial aims to compare the efficacy of a digital brief behavioural therapy for insomnia (dBBTi) against online sleep health education on insomnia symptom severity in older adults aged 60 years and over. The trial will be totally online with participants recruited from the community across Australia.

DETAILED DESCRIPTION:
Insomnia is a highly prevalent sleep disorder affecting up to 10% of the adult population and reports of over 40% in the older population. Current insomnia treatments focus heavily on symptom management with cognitive behavioural therapy for insomnia (CBTi), in both digital and face-to-face form as the recommended first-line treatment. Despite the strong evidence for digital CBTi, there are a lack of data related to older people and whether digital brief behavioural therapy is efficacious in this population.

The investigators will conduct a fully online study comparing 6-weeks of digital brief behavioural therapy for insomnia (dBBTi) against online sleep health education. Participants will be recruited, screened and determined eligibility and consent will be conducted online. Thereafter, participants will be randomly allocated to either dBBTi delivered via a mobile application called SleepFix or wait-listed control. The SleepFix app delivers sleep restriction therapy using a 4 stage approach to improve sleep efficiency. The control will consist of 3 online sleep health education modules provided bi-weekly with information about sleep and sleep hygiene without any specific insomnia therapy. Participants will be recruited using social media and directed to a website to determine eligibility and then provided access to either the dBBTi (SleepFix) or the control with a link to the first online module.

At baseline, all participants will complete self-reported measures of insomnia, sleep, fatigue, sleepiness , anxiety, depression, quality of life, cognition and digital health literacy. These will be repeated at follow-up at weeks 8, 16 and 26.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged ≥ 60 years
2. Able to give informed online consent
3. Insomnia Severity Index ≥ 10, including a score of 3 in at least one of the first three items (nocturnal symptoms).
4. English fluency
5. Access to a smartphone and willingness/proficiency to use a mobile app

Exclusion Criteria:

1. Shift-workers
2. Travel to a destination with >2 hours time-difference (within 30-days)
3. Serious medical and/or psychiatric illnesses/disorders or self-harm risk (Patient Health Questionnaire-9, item 9, 1+ score of risk of suicidal ideation)
4. Diagnosed sleep disorders other than insomnia
5. Regular sleep medications or sleep devices (>2 times a week over last 6 months)
6. Currently receiving or previously received (within the last 12 months) psychotherapy for insomnia including Cognitive Behavioural Therapy (CBT).
7. Drive for work/operate heavy machinery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in insomnia symptom severity | Change score from baseline at 8 weeks
  Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 4) regarding symptoms over the past 2 weeks. Scores range from 0-28 with higher scores indicating greater insomnia symptom severity.

SECONDARY OUTCOMES:
Change in subjective sleep quality | Change score from baseline at 8 weeks
  Subjective sleep quality will be determined from the Pittsburgh Sleep Quality Index Score (PSQI) - a 19-item questionnaire with seven component scores derived from the responses, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0-21) where a score of 5 or more indicates poor sleep quality.
Change in sleep onset latency | Change score from baseline at 8 weeks
  Sleep onset latency will be determined from the Pittsburgh Sleep Quality Index Score (PSQI) - a 19-item questionnaire with a total score range of 0 to 21 with scores greater than 5 indicating poor sleep quality. A single item will be used to assess sleep onset latency over the last 2 weeks.
Change in wake after sleep onset | Change score from baseline at 8 weeks
  Wake after sleep onset will be determined from the Pittsburgh Sleep Quality Index Score (PSQI) - a 19-item questionnaire with a total score range of 0 to 21 with scores greater than 5 indicating poor sleep quality. A single item will be used to assess wake after sleep onset over the last 2 weeks.
Change in total sleep time | Change score from baseline at 8 weeks
  Total sleep time will be determined from the Pittsburgh Sleep Quality Index Score (PSQI) - a 19-item questionnaire with a total score range of 0 to 21 with scores greater than 5 indicating poor sleep quality. A single item will be used to assess total sleep time over the last 2 weeks.
Change in fatigue | Change score from baseline at 8 weeks
  The Flinders Fatigue Scale (FFS) is a 7-item self-reported instrument designed to measure the level of subjective daytime fatigue experienced over the previous two weeks. 6-items consist of a 5-point Likert type scale ranging from "not at all" = 0 to "extremely" = 4. Item 5 uses a multiple-item checklist and is scored as a sum. All items are summed with total scores ranging from 0-31 with higher scores reflecting greater fatigue.
Change in daytime sleepiness | Change score from baseline at 8 weeks
  The Epworth Sleepiness Scale (ESS) is an 8-item self-reported questionnaire that provides a rating of general sleepiness over the last 2 weeks using a 4-point likert scale from "would never dose" = 0 to "high chance of dozing" = 3. All items are summed with total scores ranging from 0-26 where scores >10 indicating above-average daytime sleepiness.
Change in quality of Life | Change score from baseline at 8 weeks
  The EuroQol five-dimensional (EQ-5D) is a self-reported questionnaire which assesses 5 dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression and overall health. The 5 dimensions range from "1 = indicating no problem" - "5 = indicating unable to/extreme problems" and the overall score from 0 (worst health state imaginable) to 100 (best health state imaginable).
Change in depressive symptoms | Change score from baseline at 8 weeks
  The Patient Health Questionnaire-9 is a 9-item self-reported measure of depressive symptoms over the past 2 weeks. Scores for each question (Likert type scale "not at all" = 0 to "nearly every day" = 3) sum to a total score out of 27 with higher scores reflecting severe depressive symptoms.
Change in anxiety | Change score from baseline at 8 weeks
  The General Anxiety Disorder-7 (GAD-7) is a 7-item self-administered scale used to assess the severity of generalised anxiety over the previous 2 weeks. It consists of a three-point Likert type scale for each item (ranging from "not at all" = 0 to "nearly every day" = 3). All items are summed with total scores ranging from 0-21 where 5, 10 and 15 indicate the cut-off scores for mild, moderate and severe anxiety, respectively.
Change in self-reported cognition | Change score from baseline at 8 weeks
  The British Columbia Cognitive Complaints Inventory (BC-CCI) is a 6-item tool to assess self-perceived cognition. It explores any perceived problems associated with cognition, memory, expressing thoughts, word finding, slow thinking, and difficulty solving problems in reflection of the last 7 days. Answers for each question range from 0 (= "not at all") to 3 (= "Very much"). Scores are summed to a total out of 18 that reflects the cognitive complaint severity.
Engagement | Baseline, week 8
  To determine if there is a relationship between therapeutic outcome (Insomnia Severity Index, ISI) and engagement (number of in-app sleep diary entries for study completers)
The effect of baseline digital health literacy on therapy efficacy | Baseline, week 8
  Digital health literacy will be assessed using the eHEALS Literacy Scale (eHEALS) which is an 8-item, 5-point Likert-type questionnaire that measures a participant's perception of, and ability toward electronic health information. Responses range from "strongly disagree" =1, to "strongly agree" = 5. Total scores are summed to range from 8 to 40 where lower scores indicate lower self-reported digital health literacy.
  The moderating effect of the baseline digital health literacy on therapeutic outcomes (ISI scores) and engagement (number of daily sleep diary entries) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Grunstein, MD, PhD, Principal Investigator — Woolcock Institute of Medical Research; Christopher Gordon, PhD, Principal Investigator — University of Sydney
Locations (1):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data may be made available upon the Principal investigator's agreement with an amendment required to the approving ethics board.
Supporting Information: Study Protocol, ICF
Time Frame: The study data will be available following all analyses.
Access Criteria: Contact the Coordinating Principal Investigator for access to data.

REFERENCES:
- See also: Woolcock Institute of Medical Research — https://www.woolcock.org.au/
- See also: Faculty of Medicine and Health, The University of Sydney — https://www.sydney.edu.au/medicine-health/